CLINICAL TRIAL: NCT03954860
Title: Effect of no Drainage Tube on Blood Loss and Recovery After High Tibial Osteotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019041
Record Dates: First submitted 2019-05-06; First posted 2019-05-17 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2019-05

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Drainage (Experimental): The preoperative dose of tranexamic acid was calculated according to 20 mg / kg body weight, 100 ml of tranexamic acid sodium chloride solution was dripped 30 minutes before operation, and 30 ml saline containing 2 g tranexamic acid was applied to the local area before loosening the tourniquet.Postoperative intravenous drip of 100 ML sodium chloride solution containing 20 mg / kg tranexamic acid. No drainage tube was placed after operation.
  Interventions: Drug: Tranexamic Acid; Drug: Sodium Chloride 0.9%
- Drainage (Active Comparator): The preoperative dose of tranexamic acid was calculated according to 20 mg / kg body weight, 100 ml of tranexamic acid sodium chloride solution was dripped 30 minutes before operation, and 30 ml saline containing 2 g tranexamic acid was applied to the local area before loosening the tourniquet.Postoperative intravenous drip of 100 ML sodium chloride solution containing 20 mg / kg tranexamic acid. Drainage tube should be placed after operation.
  Interventions: Other: Drainage Tube; Drug: Tranexamic Acid; Drug: Sodium Chloride 0.9%

INTERVENTIONS:
Other: Drainage Tube — The drainage tube drainage to guide the pus, blood and liquid accumulated between human tissues or in body cavity outside the body of High tibial osteotomy'patients.
  Arms: Drainage
Drug: Tranexamic Acid — Tranexamic acid (TXA) is an anti-fibrinolytic drugcan，which can increase the stability of fibrin clots and achieve hemostasis for High tibial osteotomy'patients.
  Other Names: TXA
Drug: Sodium Chloride 0.9% — Sodium Chloride 0.9% is a solution of sodium chloride, which has the same osmotic pressure as animal or human plasma in physiological experiments or clinics, and can be used to dilute Tranexamic Acid .
  Other Names: sodium chloride solution

SUMMARY:
The objective of this study was to evaluate the safety and efficacy of topical combined with intravenous tranexamic acid for high tibial osteotomy without placement of a drainage tube The clinical scores of patients and their possible risks were tracked. The investigators hypothesized that a combination of tranexamic acid and no drainage tube could reduce blood loss and facilitate early recovery. The implementation of the study will provide a new perioperative blood loss control program for High Tibial Osteotomy, reduce the cost of hospitalization, promote patients to get out of bed early, reduce the number of days in hospital.

DETAILED DESCRIPTION:
The condition of the patients was evaluated, and the total length of both lower limbs, anteroposterior position of knee and Mri of knee were included. The preoperative dose of tranexamic acid was calculated according to body weight of 20 mg / kg, 100 ml of tranexamic acid sodium chloride solution was dripped 30 minutes before operation, and after incision closure, 30 ml of normal saline solution containing 2 g of tranexamic acid was injected through drainage tube or subcutaneously. Postoperative intravenous drip of 100 ML sodium chloride solution containing 20 mg / kg tranexamic acid. Arthroscopy was first used to further confirm the cartilage defect, and a new type of lower limb alignment meter and a customized precise osteotomy template were used to perform the osteotomy according to the preoperative plan. One group was not placed drainage tube, the other group was placed drainage tube. Visual analogue pain score (Vas) and American Special Surgical Hospital (HSS) knee function score were recorded 3 month after surgery. Throughout the trial, the investigators will carefully observe and manage your complications and the outcome of your surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Simple knee medial compartment osteoarthritis High tibial osteotomy.
2. With varus deformity, medial proximal tibia angle <85°
3. Unilateral High tibial osteotomy
4. informed consent: Participants must be able to understand and voluntarily sign a written informed consent and follow the research protocol and interview process

Exclusion Criteria:

1. patients who underwent other knee surgery within 6 months
2. Preoperative combined anemia (Hb<100g/l)
3. Patients with severe cardiovascular, hepatic, renal and hematopoietic diseases
4. Patient with preoperative coagulation abnormalities 5. Patients with allergies and patients allergic to TXA.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Postoperative blood loss | The third day after operation
  Total blood loss preoperative blood volume =(preoperative hematocrit-postoperative Hematocrit) + transfusion volume.
Haemoglobin | The third day after operation
  Reactive blood loss
Hematocrit | The third day after operation
  Reactive blood loss
Hospital for special surgery knee score | postoperative 3 month
  HSS is a knee function scoring system with a full score of 100. 0 means the loss of knee function, 100 means the best knee function, and the greater the value, the better knee function.
Visual Analogue Scale Postoperative Day One | Postoperative Day One
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Visual Analogue Scale Postoperative Day Three | Postoperative Day Three
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Visual Analogue Scale Postoperative Day Five | Postoperative Day Five
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Circumference of shank Postoperative Day One | Postoperative Day One
  indirectly reflects the latent blood loss
Circumference of shank Postoperative Day Three | Postoperative Day Three
  indirectly reflects the latent blood loss
Circumference of shank Postoperative Day Five | Postoperative Day Five
  indirectly reflects the latent blood loss
Number of blood transfusions | Postoperative Day Three
  If the hemoglobin was <80 g/l, allogeneic blood was transfused, and the number of blood transfusions were recorded.0 means no blood transfusion, and the larger the number is, the more blood transfusion.The maximum number does not exceed the total number of patients
Number of Incision infection | postoperative 3 month
  The incision was red, swollen, hot and painful, and the blood routine showed that the leukocyte was increased.
Number of hematoma formation | postoperative 3 month
  After operation, the incision is swollen and has wave motion, but it is not hot or painful, and there will be blood outflow during puncture.
Number of delayed healing of the incision. | On the 14th day after operation
  On the 14th day after operation, the incision did not heal.
Volume of drainage | Postoperative Day One
  Reactive blood loss

SECONDARY OUTCOMES:
Activated partial thromboplastin time | The third day after operation
  Assessment of coagulation function in patients
Prothrombin time | The third day after operation
  Assessment of exogenous coagulation system
Concentration of D-dimer | The third day after operation
  Assessment of thrombotic diseases
Concentration of Fibrinogen | The third day after operation
  Assessment of coagulation function in patients

CONTACTS AND LOCATIONS:
Overall Officials: Peilai Liu, Ph.D, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analysed during the current study are available from the overall study officials on reasonable request.

REFERENCES:
- [Background] Kim KI, Kim HJ, Kim GB, Bae SH. Tranexamic acid is effective for blood management in open-wedge high tibial osteotomy. Orthop Traumatol Surg Res. 2018 Nov;104(7):1003-1007. doi: 10.1016/j.otsr.2018.07.019. Epub 2018 Sep 20. PMID 30245067
- [Background] Palanisamy JV, Das S, Moon KH, Kim DH, Kim TK. Intravenous Tranexamic Acid Reduces Postoperative Blood Loss After High Tibial Osteotomy. Clin Orthop Relat Res. 2018 Nov;476(11):2148-2154. doi: 10.1097/CORR.0000000000000378. PMID 29939895
- [Background] Suh DW, Kyung BS, Han SB, Cheong K, Lee WH. Efficacy of Tranexamic Acid for Hemostasis in Patients Undergoing High Tibial Osteotomy. J Knee Surg. 2018 Jan;31(1):50-55. doi: 10.1055/s-0037-1600091. Epub 2017 Mar 29. PMID 28355682
- [Background] Zhang Q, Zhang Q, Guo W, Liu Z, Cheng L, Zhu G. No need for use of drainage after minimally invasive unicompartmental knee arthroplasty: a prospective randomized, controlled trial. Arch Orthop Trauma Surg. 2015 May;135(5):709-13. doi: 10.1007/s00402-015-2192-z. Epub 2015 Mar 8. PMID 25750137
- [Background] Huang Z, Xie X, Li L, Huang Q, Ma J, Shen B, Kraus VB, Pei F. Intravenous and Topical Tranexamic Acid Alone Are Superior to Tourniquet Use for Primary Total Knee Arthroplasty: A Prospective, Randomized Controlled Trial. J Bone Joint Surg Am. 2017 Dec 20;99(24):2053-2061. doi: 10.2106/JBJS.16.01525. PMID 29257010
- [Background] Chan JJ, Cirino CM, Huang HH, Poeran J, Mazumdar M, Parsons BO, Anthony SG, Galatz LM, Cagle PJ Jr. Drain Use is Associated with Increased Odds of Blood Transfusion in Total Shoulder Arthroplasty: A Population-Based Study. Clin Orthop Relat Res. 2019 Jul;477(7):1700-1711. doi: 10.1097/CORR.0000000000000728. PMID 30985612
- [Background] Legnani C, Oriani G, Parente F, Ventura A. Reducing transfusion requirements following total knee arthroplasty: effectiveness of a double infusion of tranexamic acid. Eur Rev Med Pharmacol Sci. 2019 Mar;23(5):2253-2256. doi: 10.26355/eurrev_201903_17273. PMID 30915773
- [Background] Nishitani K, Kuriyama S, Nakamura S, Ito H, Matsuda S. A Multivariate Analysis on the Effect of No Closed Suction Drain on the Length of Hospital Stay in Total Knee Arthroplasty. Knee Surg Relat Res. 2019 Mar 1;31(1):25-30. doi: 10.5792/ksrr.18.013. PMID 30871289
- [Derived] Li S, Yang J, Watson C, Lu Q, Zhang M, Miao Z, Luo D, Liu P. Drainage relieves pain without increasing post-operative blood loss in high tibial osteotomy: a prospective randomized controlled study. Int Orthop. 2020 Jun;44(6):1037-1043. doi: 10.1007/s00264-020-04530-z. Epub 2020 Mar 14. PMID 32172314